CLINICAL TRIAL: NCT06934018
Title: Effect of Surgical Margin Width on Recurrence and Survival in Patients With Hepatic Oligometastasis of Colorectal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lu Wang, MD, PhD, MD,PhD, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2503317-21
Record Dates: First submitted 2025-04-09; First posted 2025-04-18 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Oncology; Tumor Recurrence and Metastasis
Keywords: Liver metastasis of colorectal cancer
MeSH Terms: conditions — Neoplasms; Recurrence; Neoplasm Metastasis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The surgical margin width was greater than or equal to 7mm
  Interventions: Procedure: Surgery and procedure
- Control group (Experimental): The surgical margin width was less than 7mm
  Interventions: Procedure: Surgery and procedure

INTERVENTIONS:
Procedure: Surgery and procedure — According to the "Chinese Guidelines for the Diagnosis and Comprehensive Treatment of Liver metastases of Colorectal Cancer (2023 edition)", R0 resection of metastatic tumors is satisfied, and the objective is to preserve sufficient functional liver tissue, and the surgical margin width is less than 7mm
  Arms: Control group
Procedure: Surgery and procedure — Combined with intraoperative B-ultrasound guidance, 3D reconstruction and intraoperative navigation, the surgical margin width of metastatic tumor was greater than or equal to 7mm
  Arms: Experimental group

SUMMARY:
The main objective of this study was to evaluate the effect of surgical margin width on the prognosis of patients with hepatic oligometastasis of colorectal cancer by statistical 1-year intrahepatic recurrence-free survival rate (ihRFSrate). The secondary objective of the study was to evaluate the effect of surgical margin width on long-term survival and total recurrence of colorectal cancer in patients with hepatohepatic metastasis by statistical overall survival time (OS) and relapse-free survival time (RFS), and to evaluate the safety of wide margin surgery compared with narrow margin surgery in patients with Cromitis during perioperative period.

This was a single-center, prospective, randomized controlled clinical study to evaluate the effects of surgical margin width on 1-year intrahepatic relapse-free survival, relapse-free survival time, overall survival time, and perioperative safety in patients with hepatic oligometastasis of colorectal cancer. Subjects will undergo radical resection of liver tumors and will be randomly assigned to a wide margin group (≥7mm) or narrow margin group (<7mm) using stratified randomization, stratified by primary lesion site (right colon vs left colon/rectum). The margin width was the narrowest margin distance measured in fresh specimens. After radical liver tumor resection, subjects were pretreated regularly Follow-up evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, age ≥18 years;
* ECOG Physical condition score :0-1 score;
* Liver biopsy pathologic diagnosis or clinical history combined with laboratory examination and imaging findings can be used to diagnose colorectal cancer in liver;
* The primary lesion of colorectal cancer has been resected or can be resected 4-6 weeks after hepatectomy;
* The number of liver metastases was less than or equal to 5；
* There was no extrahepatic metastases or the metastases were radically resected；
* Preoperative assessment (based on enhanced CT or MRI image AI segmentation combined with three-dimensional reconstruction of hepatic parenchymal blood vessels) enables radical (R0) resection of hepatic oligometastases, and wide surgical margin (the narrowest incisal margin of fresh specimens surgically removed is greater than or equal to 7mm) can be achieved technically, and the incisal margin width is not affected by the intrahepatic vasculature；
* Good liver reserve function (preoperative Child-Pugh grade A liver function, estimated remaining liver volume ≥30%)；
* Preoperative examinations do not show clear surgical contraindications；
* Volunteer to participate in this study and sign the informed consent；
* The compliance was good, and the family members were willing to cooperate with the follow-up；

Exclusion Criteria:

* There are still untreated extra-hepatic metastases；
* Staging hepatectomy is planned, such as PVE combined with hepatectomy, ALPPS, etc；
* The number of liver metastases before chemotherapy was more than 5；
* Complicated with portal vein tumor thrombus or hepatic vein invasion；
* Concurrent with other uncured malignancies or with other primary malignancies for less than 5 years；
* Expected survival time ≤6 months；
* Those who have a history of psychotropic substance abuse and are unable to abstain or have mental disorders；
* Have a history of immunodeficiency or other acquired or congenital immunodeficiency diseases; Or have an autoimmune disease；
* According to the study, there are serious concomitant diseases that endanger the patient's safety or interfere with the patient's completion of the study；
* Patients or family members could not understand the conditions and goals of the study；

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2026-04-07 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Intrahepatic recurrence-free survival at 1 year(ihRFS rate) | From liver tumor resection to 1 year after surgery
  Refers to the percentage of subjects in this group who received intrahepatic imaging diagnosis of recurrence or death from any cause from surgery to 1 year after surgery.

SECONDARY OUTCOMES:
Recurrence free survival time(RFS) | 12 months
  The earliest date from the date of receipt of liver tumor resection to the date of confirmation of tumor recurrence or the date of death from any cause. Regular follow-up visits were conducted until the end of the study follow-up
Overall survival time(OS) | 24 months
  Refers to the time from liver tumor resection to death from any cause, if the above criteria were not met, the date of the last evaluation was used for analysis.
Perioperative safety | Patient 90 days after hepatectomy
  In this study, the incidence of perioperative complications was calculated according to Clavien Dindo complication scoring system. At the same time, perioperative death, operative time, intraoperative blood loss, blood transfusion and other surgical safety treatment were counted

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weichselbaum RR, Hellman S. Oligometastases revisited. Nat Rev Clin Oncol. 2011 Jun;8(6):378-82. doi: 10.1038/nrclinonc.2011.44. Epub 2011 Mar 22. PMID 21423255
- [Background] Su YM, Liu W, Yan XL, Wang LJ, Liu M, Wang HW, Jin KM, Bao Q, Wang K, Li J, Xu D, Xing BC. Five-year survival post hepatectomy for colorectal liver metastases in a real-world Chinese cohort: Recurrence patterns and prediction for potential cure. Cancer Med. 2023 Apr;12(8):9559-9569. doi: 10.1002/cam4.5732. Epub 2023 Feb 27. PMID 36846977
- [Background] Laroche S, Scatton O, Charlotte F, Bachet JB, Lim C, Fuks D, Goumard C. Prognosis of a Heterogeneous TRG Pathological Response to Neoadjuvant Chemotherapy in Patients who Undergo Resection for Colorectal Liver Metastases. Ann Surg Oncol. 2024 Jul;31(7):4436-4444. doi: 10.1245/s10434-024-15196-x. Epub 2024 Mar 28. PMID 38549003
- [Background] Guckenberger M, Lievens Y, Bouma AB, Collette L, Dekker A, deSouza NM, Dingemans AC, Fournier B, Hurkmans C, Lecouvet FE, Meattini I, Mendez Romero A, Ricardi U, Russell NS, Schanne DH, Scorsetti M, Tombal B, Verellen D, Verfaillie C, Ost P. Characterisation and classification of oligometastatic disease: a European Society for Radiotherapy and Oncology and European Organisation for Research and Treatment of Cancer consensus recommendation. Lancet Oncol. 2020 Jan;21(1):e18-e28. doi: 10.1016/S1470-2045(19)30718-1. PMID 31908301